CLINICAL TRIAL: NCT04565730
Title: The Effect of Different Anesthesia Methods on Development of Postnatal Depression After Cesarean Delivery: a Prospective Study
Brief Title: Different Anesthesia Methods on Development of Postnatal Depression After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol Hospital 16
Record Dates: First submitted 2020-09-16; First posted 2020-09-25 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy Related
Keywords: Anesthesia; Postnatal depression; Cesarean delivery
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is general anesthesia group. The second one is spinal anesthesia group
Who Masked: Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup I= General anesthesia group (Active Comparator): After applying standard ASA monitoring; 2-2,5 mg/kg propofol, and 0,6 mg/kg rocuronium IV will be performed for general anesthesia induction, and then orotracheal intubation will be performed. The patients will be placed in the supine position. General anesthesia will be maintained with sevoflurane in the mixture of oxygen-fresh air. Controlled mechanical ventilation will be initiated with a tidal volume of 8-10 ml/kg at 12 breaths per minute (I:E ratio 1:2), a fresh gas flow rate of 2 L per min, end tidal CO2 value at 30-35 mmHg, and peak airway pressure of maximally 30 cm H2O. All patients will undergo cesarean delivery surgery with the same technique by the same surgical team.
  Interventions: Other: Grup I= General anesthesia group
- Grup II= Spinal anesthesia group (Active Comparator): A standardized spinal anesthesia will administrated to the patients. After skin disinfection, 25G needle will used for puncture at the level of L2-L3 or L3-L4. After observing the cerebrospinal fluid, 15 mg bupivacaine (marcain spinal heavy) will be administered into the subarachnoid space. The level of anesthesia below T6 will be controlled.
  Interventions: Other: Grup II= Spinal anesthesia group

INTERVENTIONS:
Other: Grup I= General anesthesia group — Preoperative and postoperative evaluation Pre-operative data will be collected 1 to 2 hrs before operation. Preoperative anxiety level will be assessed by the Hospital Anxiety and Depression Scale (HADS) and Amsterdam Preoperative Anxiety and Information Scale.
  Patients will be asked to complete the Edinburgh Postnatal Depression Scale (EPDS) on the morning of discharge, 1 months and 3 months days after delivery. An online survey will be conducted post-Cesarean delivery to investigate the primary outcome of PND using EPDS, and those will not complete the online survey received phone calls to conduct the follow-up surveys.
  Arms: Grup I= General anesthesia group
Other: Grup II= Spinal anesthesia group — Preoperative and postoperative evaluation Pre-operative data will be collected 1 to 2 hrs before operation. Preoperative anxiety level will be assessed by the Hospital Anxiety and Depression Scale (HADS) and Amsterdam Preoperative Anxiety and Information Scale.
  Patients will be asked to complete the Edinburgh Postnatal Depression Scale (EPDS) on the morning of discharge, 1 months and 3 months days after delivery. An online survey will be conducted post-Cesarean delivery to investigate the primary outcome of PND using EPDS, and those will not complete the online survey received phone calls to conduct the follow-up surveys.
  Arms: Grup II= Spinal anesthesia group

SUMMARY:
Childbirth is one of the most painful experiences for a woman. Labor and period of pregnancy is associated with an increased risk of psychiatric disorders for a woman. The demands of pregnancy and childbirth make patients vulnerable to psychiatric disorders such as postpartum depression (PPD), anxiety, and stress disorders. Women with postpartum psychiatric disorders have high mortality rates. The most common postpartum psychiatric disorder is PPD. PPD occurs any time in pregnancy or in the first four weeks after delivery. It may lead to complications such as emotional lability in the mother. This situation may also effect the child.

DETAILED DESCRIPTION:
Childbirth is one of the most painful experiences for a woman. Labor and period of pregnancy is associated with an increased risk of psychiatric disorders for a woman. The demands of pregnancy and childbirth make patients vulnerable to psychiatric disorders such as postpartum depression (PPD), anxiety, and stress disorders. Women with postpartum psychiatric disorders have high mortality rates. The most common postpartum psychiatric disorder is PPD. PPD occurs any time in pregnancy or in the first four weeks after delivery. It may lead to complications such as emotional lability in the mother. This situation may also effect the child.

Postpartum depression (PD) has become the most frequent complication of childbirth. Its prevalence has been estimated as 10%-15% and its formation is affected by several factors such as lack of social support, previous history of depression, and personal vulnerability. There are several studies about PD in the literature, some discuss about the relation of pain and PD, some discuss about the relation of epidural anesthesia and PD. However, there is no study that compares different anesthesia methods (general anesthesia vs spinal anesthesia) on development of postnatal depression after cesarean delivery.

The aim of this study is to compare the different anesthesia methods (general anesthesia vs spinal anesthesia) on development of postnatal depression after cesarean delivery. The secondary aim is to decrease the ratio of postnatal depression after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-50 years old
* 36 gestational weeks or more,
* American Society of Anesthesiologists' (ASA) I and II
* Able to communicate

Exclusion Criteria:

* history of bipolar or psychotic disorder
* suicidal state
* Chronic pain syndrome
* Intraoperative complication
* drug and/or alcohol abuse
* who did not want to participate
* emergency cases
* unable to communicate in Turkish

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients
Enrollment: 200 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Development of postnatal depression | Change from baseline Edinburgh Postnatal Depression Scale (EPDS) before discharge, 1 months and 3 months days after delivery.
  The aim of this study is to compare the different anesthesia methods (general anesthesia vs spinal anesthesia) on development of postnatal depression after cesarean delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Munro A, MacCormick H, Sabharwal A, George RB. Pharmacologic labour analgesia and its relationship to postpartum psychiatric disorders: a scoping review. Can J Anaesth. 2020 May;67(5):588-604. doi: 10.1007/s12630-020-01587-7. Epub 2020 Feb 4. PMID 32020416
- [Background] Kaya L, Cigdem Z. The relationship between mode of delivery and postpartum depression. J Educ Health Promot. 2019 Jan 29;8:5. doi: 10.4103/jehp.jehp_97_18. eCollection 2019. PMID 30815476
- [Background] Chan CL, Tan CW, Chan JJI, Sultana R, Chua TE, Chen HY, Sia ATH, Sng BL. Factors Associated with the Development of Postnatal Depression After Cesarean Delivery: A Prospective Study. Neuropsychiatr Dis Treat. 2020 Mar 12;16:715-727. doi: 10.2147/NDT.S241984. eCollection 2020. PMID 32210566
- [Background] Zanardo V, Giliberti L, Volpe F, Parotto M, de Luca F, Straface G. Cohort study of the depression, anxiety, and anhedonia components of the Edinburgh Postnatal Depression Scale after delivery. Int J Gynaecol Obstet. 2017 Jun;137(3):277-281. doi: 10.1002/ijgo.12138. Epub 2017 Mar 22. PMID 28258970
- [Background] Yu HY, Wang SY, Quan CX, Fang C, Luo SC, Li DY, Zhen SS, Ma JH, Duan KM. Dexmedetomidine Alleviates Postpartum Depressive Symptoms following Cesarean Section in Chinese Women: A Randomized Placebo-Controlled Study. Pharmacotherapy. 2019 Oct;39(10):994-1004. doi: 10.1002/phar.2320. Epub 2019 Sep 15. PMID 31411762